CLINICAL TRIAL: NCT01395420
Title: A Phase I Open-Label, 2-Part, 3-Cohort, Single-Centre Study to Assess the Concentration of Avibactam and Ceftazidime in Epithelial Lining Fluid (ELF) and Plasma Using at Least Two Different Dosing Regimens in Healthy Volunteers
Brief Title: Study to Assess the Concentration of Avibactam and Ceftazidime in Epithelial Lining Fluid and Plasma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D4280C00009
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Phase 1; open label; healthy male and female (post menopausal) volunteers; Pharmacokinetics; CAZ104; Avibactam; Ceftazidime; open label, at least 2 different regimens, concentration of investigational product (IP), CAZ104, Avibactam, Ceftazidime, Cmax, tmax
MeSH Terms: interventions — Ceftazidime; avibactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CAZ104 (2000mg Ceftazidime/500mg Avibactam)
  Interventions: Drug: CAZ104
- 2 (Experimental): CAZ104 (3000mg Ceftazidime/1000mg Avibactam)
  Interventions: Drug: CAZ104

INTERVENTIONS:
Drug: CAZ104 — IV Infusion
  Other Names: CAZ104 (2000mg Ceftazidime/500mg Avibactam)
  Arms: 1
Drug: CAZ104 — IV Infusion
  Other Names: CAZ104 (3000mg Ceftazidime/1000mg Avibactam)
  Arms: 2

SUMMARY:
This is an open-label study divided in 2 parts and 3 cohorts to determine the concentration of Avibactam and Ceftazidime in the lining of the lungs and the blood.

DETAILED DESCRIPTION:
A Phase I Open-Label, 2-Part, 3-Cohort, Single-Centre Study to Assess the Concentration of Avibactam and Ceftazidime in Epithelial Lining Fluid and Plasma Using at Least Two Different Dosing Regimens in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male and female subjects with veins suitable for cannulation or repeated venepuncture; female subjects must be postmenopausal or surgically sterile. Female subjects must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-child-bearing potential
* Male subjects should be willing to use barrier contraception ie, condoms, from dosing to 3 months after dosing with the IP
* Have a body mass index (BMI) between 19 and 30 kg/m2
* As judged by the Investigator, all the subjects must be able to understand and be willing to comply with study procedures, restrictions and requirements

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder (including a history of chronic respiratory disease eg, asthma, chronic obstructive pulmonary disease [COPD], cystic fibrosis or interstitial lung disease) which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Known allergy to lidocaine/lignocaine, midazolam, alfentanyl or other topical anaesthetics/sedatives in similar classes to these agents
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IP
* Any clinically significant abnormalities in physical examination, lung function test, ECG, clinical chemistry, haematology, coagulation screen, or urinalysis results as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To measure and compare the concentration of Avibactam and Ceftazidime in ELF and plasma | at several timepoints from pre-dose up to 5 days post dose (Part 2)
  To measure and compare the concentration of Avibactam and Ceftazidime in ELF and plasma by assessment of maximum concentration (Cmax), time to Cmax (tmax), area under the concentration time curve during a dosing interval t (AUCτ), terminal half life (t½λz) in plasma and ELF, plasma clearance (CL), volume of distribution at steady state (Vss) and at the terminal phase (Vz) in plasma, ratio of Cmax in ELF over Cmax in plasma and ratio of AUCτ in ELF over AUCτ in plasma.

SECONDARY OUTCOMES:
To evaluate safety and tolerability of Avibactam and Ceftazidime | at several timepoints from pre-dose up to 5 days post dose
  To evaluate safety and tolerability of Avibactam and Ceftazidime by assessment of adverse events (AEs), physical examinations, vital signs, 12 lead electrocardiograms (ECGs), Pulse oximetry and safety laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newell, MD, Study Director — AstraZeneca; Leonard Siew, MBCHB, MRCP(UK), Principal Investigator — Quintiles Phase I unit London; Mirjana Kujacic, MD, Study Chair — AstraZeneca
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Background] Nicolau DP, Siew L, Armstrong J, Li J, Edeki T, Learoyd M, Das S. Phase 1 study assessing the steady-state concentration of ceftazidime and avibactam in plasma and epithelial lining fluid following two dosing regimens. J Antimicrob Chemother. 2015 Oct;70(10):2862-9. doi: 10.1093/jac/dkv170. Epub 2015 Jul 1. PMID 26133566
- See also: Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1455&filename=D4280C00009%20Clinical%20Study%20009%20Protocol%20Redaction.pdf